CLINICAL TRIAL: NCT04501900
Title: The Standard Versus Prolonged Dual Antiplatelet Therapy After the XINSORB Bioresorbable Scaffold Implantation Trial
Brief Title: The 3 Years vs 1 Year DAPT After XINSORB BRS Implantation
Acronym: SPARTA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS20200804
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Clopidogrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prolonged DAPT group (Active Comparator)
  Interventions: Drug: Clopidogrel
- standard DAPT group (No Intervention)

INTERVENTIONS:
Drug: Clopidogrel — Study subjects diagnosed as stable, unstable ischemic coronary disease or myocardial infarction planning to undergo percutaneous coronary intervention (PCI) and no contradiction to prolonged DAPT are eligible for this trial. All subjects will provide written informed consent to participate. Subjects will be enrolled into the study before or within 24 hours after the index procedure. Subjects will be randomized to either discontinue P2Y12 inhibitor (clopidogrel or ticagrelor) (12 months total) or receive P2Y12 inhibitor for an additional 24 months (36 months total). Aspirin will be maintained in the entire study and can be replaced by cilostazol or indobufen if subjects are intolerant. Dosage of antiplatelet drugs will be according to local standard of practice. Subjects will be treated with XINSORB BRS only.
  Arms: prolonged DAPT group

SUMMARY:
The aim of the SPARTA trial is to clarify the impact of extending DAPT beyond 1 year after XINSORB BRS implantation by investigating the balance of risk and benefit in a broad population of treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with XINSORB BRS implantation, then treated with DAPT for 12 months
2. Written informed consent from the subjects
3. Qualified candidates for coronary bypass surgery
4. Lesions with reference vessel diameter 2.75 to 3.5 mm

Exclusion Criteria:

1. Age ≤ 18 years
2. Cardiogenetic shock
3. Chronic heart failure with a left ventricular ejection fraction ≤ 30%
4. Oral anticoagulation therapy
5. Known allergy or intolerance to the study medications
6. Malignancies and other comorbid conditions with a life expectancy less than 5 years
7. Subjects treated with both BRS and DES during the index procedure
8. Pregnant wowen
9. Planned staged PCI
10. Contemporaneous enrollment in a different clinical trial
11. Any revascularization within 1 year
12. Planned surgery necessitating discontinuation of antiplatelet therapy within 36 months after enrollment
13. Unprotected left main artery
14. Lesions located at the ostium of the main coronary artery
15. bifurcation lesions (Medina 1,1,1) planning to be treated with two stents strategy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2106 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
MACE | 3 years
  The incidence of a composite endpoint, including all-cause death, any myocardial infarction (MI), and all revascularization
BARC type 3, 4, and 5 bleeding events | 3 years

REFERENCES:
- [Derived] Wu Y, Yin J, Li C, Zhang W, Shen L, Ge L, Qian J, Ge J. The standard versus prolonged dual antiplatelet therapy after the XINSORB bioresorbable scaffold implantation (SPARTA) trial: study protocol for a randomized controlled trial. Trials. 2023 Jan 20;24(1):49. doi: 10.1186/s13063-022-07028-8. PMID 36670441